CLINICAL TRIAL: NCT05849987
Title: Retinitis Pigmentosa Clinical Study: Examining the Clinical Trial Journey of Retinitis Pigmentosa Patients
Brief Title: In Depth Observational Clinical Trial Of Retinitis Pigmentosa Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 92030990
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Typically, clinical research participation favors a specific demographic group, and little research exists on how trial attributes affect participation. As such, this study seeks to analyze data from different demographic groups and check for recurring trends that could provide valuable insights for future retinitis pigmentosa patients.

ELIGIBILITY:
Inclusion Criteria:

* Is 18+ years old
* Confirmed diagnosis of retinitis pigmentosa
* Signed Written Informed Consent

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Participant is actively receiving study therapy in another trial
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retinitis Pigmentosa patients who are actively considering enrolling in an interventional clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of patient decides to enroll in clinical trial | 3 months
Rate of patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miura G, Sugawara T, Kawasaki Y, Tatsumi T, Nizawa T, Baba T, Hanaoka H, Yamamoto S. Clinical Trial to Evaluate Safety and Efficacy of Transdermal Electrical Stimulation on Visual Functions of Patients with Retinitis Pigmentosa. Sci Rep. 2019 Aug 12;9(1):11668. doi: 10.1038/s41598-019-48158-5. PMID 31406205
- [Background] Arslan U, Ozmert E, Demirel S, Ornek F, Sermet F. Effects of subtenon-injected autologous platelet-rich plasma on visual functions in eyes with retinitis pigmentosa: preliminary clinical results. Graefes Arch Clin Exp Ophthalmol. 2018 May;256(5):893-908. doi: 10.1007/s00417-018-3953-5. Epub 2018 Mar 15. PMID 29546474
- [Background] Berson EL, Rosner B, Sandberg MA, Weigel-DiFranco C, Moser A, Brockhurst RJ, Hayes KC, Johnson CA, Anderson EJ, Gaudio AR, Willett WC, Schaefer EJ. Clinical trial of docosahexaenoic acid in patients with retinitis pigmentosa receiving vitamin A treatment. Arch Ophthalmol. 2004 Sep;122(9):1297-305. doi: 10.1001/archopht.122.9.1297. PMID 15364708

DOCUMENTS (1):
  • Informed Consent Form (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT05849987/ICF_000.pdf